CLINICAL TRIAL: NCT03559283
Title: Using Functional Near-infrared Spectroscopy (fNIRS) in the Evaluation of Cognitive-motor Interference in Post-stroke Patients
Brief Title: fNIRS in the Evaluation of Cognitive-motor Interference in Post-stroke Patients
Acronym: ICM-AVC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 87RC17_0074 (ICM AVC)
Record Dates: First submitted 2018-06-06; First posted 2018-06-18 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2019-06

CONDITIONS: D020521
Keywords: stroke, dual-task, gait parameters, fNIRS
MeSH Terms: conditions — Stroke | interventions — Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Walking and Record Cortical Activity (Experimental): A sensor placement will be performed on the patient's forehead to record brain activity when walking, when performing a mental task, and when performing both tasks at the same time. In parallel, walking will be on a carpet that will record the spatio-temporal parameters of walking.
  Interventions: Diagnostic Test: Walking and Record Cortical Activity

INTERVENTIONS:
Diagnostic Test: Walking and Record Cortical Activity — The cortical activity of each patient is recorded by NIRS under the following conditions:
  * Simple task : The patient walks on an electronic walking track (GAITRite system) over 10 meters. The data collected are the spatio-temporal parameters of walking.
  * Cognitive task alone : two conditions of the n-back test (1-back and 2-back) to study neural activities related to working memory. The duration of realization will be 30 seconds by condition and we retain the number of errors realized.
  * Double Task : Achievement of the motor task (10-meter walk) is performed at the same time as a "weak" cognitive task (1-back) and a "high" cognitive task (2-back). The spatio-temporal parameters and the number of errors are collected by the observer.

SUMMARY:
This study evaluates cognitive-motor interference in stroke patients who is responsible an alteration of spatio-temporal gait parameters. It's proved in the literature but the underlying pathophysiological mechanisms remain poorly understood. fNIRS is a functional imaging technique that evaluates this interference under optimal conditions. The purpose of this study is to evaluate the hemodynamic activity of the CPF in walking post-stroke patients under different DT conditions.

DETAILED DESCRIPTION:
Walking is a motor task that involves cognitive functions. The parameters of walking and brain activity are modified in situations requiring significant attentional and cognitive demand. fNIRS is an interesting functional neuroimaging technique for studying cortical activity when performing a Dual Task (DT). To our knowledge, no studies have examined cerebral oxygenation levels in post-stroke patients based on different cognitive loads during walking. Understanding cognitive contributions in a dual-task walking situation is necessary to providing targeted interventions and preventing falls.

Patients included in the study will be evaluated in single cognitive task, with two levels of difficulty, single walking motor task, and dual task with two levels of cognitive difficulty. The fNIRS will record the hemodynamic activity of the prefrontal cortex for the cognitive slope and the GAITRite will record the walking parameters.

ELIGIBILITY:
Inclusion Criteria:

* patient between 55 and 75 years old
* First stroke
* ischemic sylvian or hemorrhagic lobar deep respecting the frontal lobe, subacute phase (J15-J90),
* patient walking 10 meters.

Exclusion Criteria:

* Heminegligencia,
* a history of neurological pathologies, orthopedic pathologies, aphasia, cognitive disorders preceding stroke (dementia, head trauma), acute cardiovascular or respiratory pathologies.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

PRIMARY OUTCOMES:
Cost of the Double Task | Day of the Inclusion
  the double task (DT) cost measured by the average difference in magnitude of hemodynamic responses in HbO2 at the CPF level obtained by the fNIRS between the DT high and low cognitive load.

SECONDARY OUTCOMES:
Impact of the double task on spatio-temporal parameters of walking and on cognition | Day of the Inclusion
  Spatio-temporal parameters (walking speed, walking time, cadence, pitch length and pitch variability) of walking, measured on GAITRite as a function of the cognitive load of the Double Task (DT)
Evaluate the asymmetry of cerebral activation in different walking conditions | Day of the Inclusion
  Measurement of the mean difference of hemodynamic HbO2 activation of the CPF between the lesional side and the contralateral side by fNIRS as a function of the cognitive load in Double Task (DT).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Limoges, France

IPD SHARING:
Plan to Share IPD: No